CLINICAL TRIAL: NCT00497991
Title: A Phase I/II, Open Label, Multi-centre Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of AZD1152 in Patients With Acute Myeloid Leukaemia.
Brief Title: Safety, Tolerability, PK and Efficacy of AZD1152 in Patients With Relapsed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1531C00007; EUDRACT number 2005-004243-65
Record Dates: First submitted 2007-07-05; First posted 2007-07-09 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Myeloid Leukemia
Keywords: AML; phase I/II; AZD1152; Acute Myeloid Leukaemia
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia, Myeloid, Acute | interventions — 2-((3-((4-((5-(2-((3-fluorophenyl)amino)-2-oxoethyl)-1H-pyrazol-3-yl)amino)quinazolin-7-yl)oxy)propyl)(ethyl)amino)ethyl dihydrogen phosphate

INTERVENTIONS:
Drug: AZD1152

SUMMARY:
The purpose of this study is to assess safety and tolerability of multiple ascending doses of AZD1152 and to assess effect of AZD1152 on the rate of complete remission in patients with relapsed acute myeloid leukaemia.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory AML for which no standard therapies are anticipated to result in durable remission
* Newly diagnosed AML who are not considered suitable for other treatments.

Exclusion Criteria:

* Previous myeloablative therapy allogeneic bone marrow or stem cell transplantation, radiotherapy or chemotherapy within 4 weeks of first dose.
* Participation in any other trial with an investigational product within the previous 30 days
* Other active malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-05; Primary Completion 2009-10 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of multiple ascending doses AZD1152 in patients with AML by assessment of AEs, vital signs, ECG parameters, clinical chemistry, haematology (including clotting parameters) and urinalysis. | Assessed at each visit
To determine the rate of complete remission from baseline changes in bone marrow and blood myeloblast counts and recovery of normal haemopoiesis | Change from baseline

SECONDARY OUTCOMES:
To determine the pharmacokinetics, pharmacodynamics, efficacy, safety and tolerability | Assessed at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Paul Stockman, MD, Study Director — AstraZeneca; Bob Lowenberg, MD, PhD, Principal Investigator — Cancer Institute
Locations (10):
- United States (2):
  - Research Site, New York, New York
  - Research Site, Houston, Texas
- France (3):
  - Research Site, Angers
  - Research Site, Grenoble
  - Research Site, Le Chesnay
- Italy (2):
  - Research Site, Bologna
  - Research Site, Roma
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Nijmegen
  - Research Site, Rotterdam

REFERENCES:
- [Derived] Lowenberg B, Muus P, Ossenkoppele G, Rousselot P, Cahn JY, Ifrah N, Martinelli G, Amadori S, Berman E, Sonneveld P, Jongen-Lavrencic M, Rigaudeau S, Stockman P, Goudie A, Faderl S, Jabbour E, Kantarjian H. Phase 1/2 study to assess the safety, efficacy, and pharmacokinetics of barasertib (AZD1152) in patients with advanced acute myeloid leukemia. Blood. 2011 Dec 1;118(23):6030-6. doi: 10.1182/blood-2011-07-366930. Epub 2011 Oct 5. PMID 21976672